CLINICAL TRIAL: NCT00404014
Title: A Phase II Study Designed to Evaluate the Safety, Tolerability, and Effect of a Single, Rising Dose of Intravenous AL-208, Followed by a Placebo-Controlled, Double-Blind, Parallel-Group Evaluation of a Single Dose of AL-208, on Mild Cognitive Impairment Following Coronary Artery Bypass Graft Surgery.
Brief Title: Study to Evaluate Safety, Tolerability, and Effect of AL208 on Mild Cognitive Impairment Following Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL 208-201
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Mild Cognitive Impairment
Keywords: MCI following CABG surgery
MeSH Terms: conditions — Cognitive Dysfunction | interventions — davunetide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AL-208 (Active Comparator): 1 dose of 300 mg
  Interventions: Drug: AL-208
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AL-208 — 1 dose of 300 mg
  Arms: AL-208
Drug: Placebo — 1 dose of placebo
  Arms: Placebo

SUMMARY:
The primary objective is to compare mild cognitive impairment in the AL-208 group with the placebo group at 14 + - 3 days after CABG surgery

ELIGIBILITY:
Inclusion Criteria:

1. Males and females (of non-childbearing potential), 50 to 79 years of age.
2. Undergoing CABG surgery with the use of extracorporeal circulation.
3. Willing and able to complete cognitive testing.
4. Score < 16 on the Center for Epidemiological Studies in Depression scale (CES-D).
5. Score > or = 28 on the Mini-Mental State Examination (MMSE).
6. Willing and able to provide informed consent to participate in this study
7. Fluency in written and spoken English.

Exclusion Criteria:

1. Presence of any severe mental illness that could affect interpretation of efficacy data, such as schizophrenia or bipolar affective disorder; any untreated or unstable psychiatric condition including depressive disorder or anxiety disorder.
2. History of stroke or other significant neurological disorder
3. Transient ischemic attack (TIA) with ongoing cognitive sequelae
4. Chronic atrial fibrillation or uncontrolled atrial fibrillation prior to surgery
5. Myocardial infarction (MI) within the last 8 weeks and/or previous history of more than 3 MIs
6. History of liver dysfunction with ongoing sequelae (including but not limited to liver enzymes > 2.5 x upper limit or normal (ULN) at screening).
7. History of renal dysfunction with ongoing sequelae (including but not limited to creatinine value > 2.5 mg/dL at screening).
8. Known active alcohol or drug abuse.
9. Concurrent use of prescription medications known to enhance memory
10. General anesthesia (defined as anesthesia requiring intubation or ventilatory support) within 3 months prior to randomization.
11. Cardiopulmonary bypass or thoracotomy within 2 years prior to randomization.
12. Undergoing valvular repair or replacement during scheduled CABG surgery.
13. Chronic obstructive pulmonary disease (COPD) requiring oxygen therapy.
14. Decompensating congestive heart disease
15. Subjects on immunosuppressive drugs, such as azathioprine, chemotherapeutic agents, mycophenolate, monoclonal antibodies, or more than 20 mg/day prednisone, within the previous 3 months
16. Receipt of any investigational agent or device within 30 days of screening.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2006-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study was to compare mild cognitive impairment in the AL-208 group with the placebo group at 14±3 days after coronary artery bypass graft (CABG) surgery. | 14 days
  The primary objective of this study was to compare mild cognitive impairment in the AL-208 group with the placebo group at 14±3 days after coronary artery bypass graft (CABG) surgery.

SECONDARY OUTCOMES:
The safety profile of AL-208 in subjects undergoing CABG surgery | 14 days
  The safety profile of AL-208 in subjects undergoing CABG surgery
The effect of treatment with AL-208 on postoperative personality changes in subjects undergoing CABG surgery | 14 days
  The effect of treatment with AL-208 on postoperative personality changes in subjects undergoing CABG surgery
Concentration of AL-208 in plasma in subjects undergoing CABG surgery | 14 days
  Concentration of AL-208 in plasma in subjects undergoing CABG surgery

CONTACTS AND LOCATIONS:
Overall Officials: Elena Matthews, MD, Study Director — Medical Monitor on behalf of Allon Therapeutics
Locations (28):
- United States (26):
  - Physicians Clinical Research Corp., Laguna Hills, California
  - Sacramento Heart and Vascular Research Center, Sacramento, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Miami Research Associates, South Miami, Florida
  - Piedmont Hospital Research Institute, Atlanta, Georgia
  - The Atlanta Heart and Vascular Research Group, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Chicago Heart Institute and Vein Clinic, Elk Grove Village, Illinois
  - Illinois Heart and Vascular Foundation, Hindsdale, Illinois
  - Indiana/Ohio Heart Cardiothoracic and Vascular Surgeons, Fort Wayne, Indiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Cardiothoracic Associates, Flint, Michigan
  - NYU Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Carolina Cardiovascular Surgical Associates, PA, Raleigh, North Carolina
  - Memory Assessment and Research Services, Wilmington, North Carolina
  - St. Vincent Mary Medical Center, Toledo, Ohio
  - Tulsa Clinical Resesarch, LLC, Tulsa, Oklahoma
  - Consultants in Cardiovascular Diseases Inc., Erie, Pennsylvania
  - Clinical Research Solutions, PC, Knoxville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Clinical Cardiovascular Research Center, Dallas, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Cardiac and Thoracic Surgical Associates, Ltd., Mechanicsville, Virginia
  - Multicare Health Systems, Tacoma, Washington
- Canada (2):
  - London health Sciences Centre, London, Ontario
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Gozes I, Blatt J, Guz LS. Systemic davunetide provides sex-specific neuroprotection during Coronary Artery Bypass Grafting (CABG). Transl Psychiatry. 2025 Oct 31;15(1):454. doi: 10.1038/s41398-025-03675-y. PMID 41173865